CLINICAL TRIAL: NCT04315363
Title: Changing and Understanding Motivation to Increase Physical Activity Among Sedentary Older Adults
Brief Title: Daily Activity Study of Health: Increasing Physical Activity in Aging
Acronym: DASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Maiya Geddes, Affiliate Associate Professor, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 19-06-05; P30AG048785 (NIH)
Record Dates: First submitted 2020-02-26; First posted 2020-03-19 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Aging
Keywords: motivation
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Brain MRI and Motivational Behavioral Intervention
  Interventions: Behavioral: Motivational MRI and Behavioral Intervention
- Active control (Active Comparator): Brain MRI and Control Behavioral Intervention
  Interventions: Behavioral: Control MRI and Behavioral Intervention

INTERVENTIONS:
Behavioral: Motivational MRI and Behavioral Intervention — Motivational messaging delivered during a functional brain MRI scan and with daily messaging
  Arms: Intervention
Behavioral: Control MRI and Behavioral Intervention — Control messaging delivered during a functional brain MRI scan and with daily messaging
  Arms: Active control

SUMMARY:
In this six-week behavioral intervention, sedentary older adults will receive daily health messaging via their smart phone to better understand their daily activities and emotions. Participants undergo structural and functional brain imaging before and after the intervention along with measures of their behavioral, emotional and thinking functions.

DETAILED DESCRIPTION:
This project will obtain data on the effects of a six week intervention designed to increase subjects' motivation to increase their physical activity. Subjects will be randomized into two different conditions to examine the efficacy of self-affirmation + positive messaging versus a control group that receives negative messaging only on changes in physical activity.

We will also examine whether any differential physical activity or structured exercise engendered in the two groups is maintained at 3 months post-intervention.

Secondary outcome measures will include a battery of cognitive, psychosocial, and neuroimaging measures that are designed to explicate the mechanisms that underlie motivation effects for physical activity in sedentary older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age range 60-95
* Not exercising more than 150 minutes of moderate/vigorous intensity per week AND sitting more than 8 hours per day
* No contraindications to MRI (if opting for MRI)
* Being able to speak English fluently
* Body Mass Index (BMI) between 20 and 40
* Normal or corrected-normal vision based on the minimal 20/20 standard
* Ambulatory without severe pain or the assistance of walking devices
* No diagnosis of a neurological disease
* Regular access to a computer with internet or smartphone

Exclusion Criteria:

* Primary care physician does not approve additional physical activity
* Inability to ambulate without assistive device
* Any unstable medical condition
* Current diagnosis of a Diagnostic and Statistical Manual of Mental Disorders (DSM-V) Axis I or II disorder including Major Depression
* History of major psychiatric illness including schizophrenia (not including general anxiety disorder or depression)
* Current treatment for cancer - except non-melanoma skin
* Neurological condition (multiple sclerosis, Parkinson's disease, dementia, mild cognitive impairment) or brain injury (traumatic or stroke)
* Current alcohol or substance abuse
* Current treatment for congestive heart failure, angina, uncontrolled arrhythmia, deep vein thrombosis or other cardiovascular event
* Myocardial infarction, coronary artery bypass grafting, angioplasty or other cardiac condition in the past year
* Not passing the Telephone Interview of Cognitive Status (TICS) as normal
* Use of any anti-psychotic, anti-depressant, anti-anxiety, and attention deficit disorder (ADD/ADHD) medications.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ai M, Morris TP, Ordway C, Quinonez E, D'Agostino F, Whitfield-Gabrieli S, Hillman CH, Pindus DM, McAuley E, Mayo N, de la Colina AN, Phillips S, Kramer AF, Geddes M. The Daily Activity Study of Health (DASH): A pilot randomized controlled trial to enhance physical activity in sedentary older adults. Contemp Clin Trials. 2021 Jul;106:106405. doi: 10.1016/j.cct.2021.106405. Epub 2021 May 1. PMID 33945886

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Brain MRI and Motivational Behavioral Intervention
  Behavioral Intervention: Motivational messaging (self affirmation on highest ranked value and positively framed messages) delivered as daily messages, and due to the pandemic, a functional brain MRI scan at baseline was optional
- Active Control: Brain MRI and Control Behavioral Intervention
  Control Behavioral Intervention: Control motivational messaging (self affirmation on lowest ranked value and negatively framed messages) delivered as daily messages, and due to the pandemic, a functional brain MRI scan at baseline was optional
Period: Overall Study
Arm/Group | Intervention | Active Control
Started | 21 | 19
Completed | 21 | 17
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Active Control | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (5.4) | 68.4 (5.0) | 68.7 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 6 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 7 | 0 | 7
  White/Caucasian | 12 | 17 | 29
  Asian/Pacific Islander | 2 | 1 | 3
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40
education [Mean (Standard Deviation); unit: years] | 16.6 (3.6) | 16.0 (3.6) | 16.3 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sedentary Behavior (Average Hour/Day)
Description: This metric quantifies the change in the average amount of time spent sedentary each day in hours, from the baseline period to the 6-week follow-up period. It is a marker of time spent inactive.
Time Frame: Baseline; 6-week
Population: The number of average daily hours spent sedentary after the intervention compared to the pre-intervention baseline.
Measure: Mean (Standard Deviation); unit: Change in average daily hours
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 21 | 17
Change in average daily hours | -0.11 (1.62) | 0.05 (1.61)
Statistical Analysis 1: Comparison: Intervention vs Active Control; Test type: Equivalence — Two by two Mixed Analysis of Variance (ANOVA) models (i.e., within-subject effect: pre- and post- intervention * between-subject effect: intervention and control group) were estimated to investigate the primary outcome changes (i.e., sedentary time) before and after the intervention; p = 0.8, ANOVA

2. Secondary Outcome: Change in Moderate-to-Vigorous Physical Activity
Description: This measure focuses on the change in average moderate-to-vigorous physical activity (MVPA) daily minutes after the intervention compared to the pre-intervention average MVPA baseline.
Time Frame: Baseline; 6-week
Population: The change in average number of daily minutes spent in moderate-to-vigorous physical activity after the intervention compared to the pre-intervention baseline.
Measure: Mean (Standard Deviation); unit: Change in minutes daily
Arm/Group | Intervention | Active Control
Number analyzed (Participants) | 21 | 19
Change in minutes daily | -0.17 (1.09) | 0.14 (0.41)
Statistical Analysis 1: Comparison: Intervention vs Active Control; Test type: Equivalence — Two by two Mixed Analysis of Variance (ANOVA) models (i.e., within-subject effect: pre- and post- intervention * between-subject effect: intervention and control group) were estimated to investigate the secondary outcome changes (i.e., moderate-to-vigorous physical activity) before and after the intervention; p = 0.35, ANOVA

ADVERSE EVENTS:
Time Frame: Duration of the study (6-week intervention and baseline visit)
Arm/Group | Intervention | Active Control
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

LIMITATIONS AND CAVEATS:
Given that the trial was conducted during lockdowns due to the COVID-19 pandemic, the original brain imaging MRI outcomes were modified. Intervention delivery was remote due to in-person data collection restrictions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT04315363/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT04315363/SAP_001.pdf